CLINICAL TRIAL: NCT00001026
Title: A Phase I, Multicenter, Randomized Trial to Evaluate the Safety and Immunogenicity of a Recombinant Vaccinia-HIV Envelope Vaccine (HIVAC-1e) in Combination With a Panel of Subunit Recombinant HIV Envelope Vaccines in Vaccinia-Naive Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 010; 10555 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; HIV Envelope Protein gp160; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — HIVAC-1e

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)
Biological: rgp120/HIV-1IIIB
Biological: rgp120/HIV-1MN
Biological: rgp120/HIV-1 SF-2
Biological: HIVAC-1e

SUMMARY:
Primary: To determine whether combination vaccination, i.e., priming with a vaccinia recombinant-containing HIV envelope (HIVAC-1e) followed by boosting with a recombinant subunit envelope protein (gp160 or gp120), provides enhanced immunogenicity compared to subunit vaccination with the individual recombinant envelope proteins only. To compare the relative immunogenicity of a panel of HIV envelope subunit vaccines when administered as boosters following recombinant HIV-vaccinia priming. To evaluate the relative immunogenicity of one versus two doses of recombinant HIV-vaccinia prior to the subunit protein boost.

Secondary: To examine the safety of administering the individual subunit vaccines in combination with the HIV envelope vaccinia recombinant, and to extend the population to whom these proteins have been administered.

Previous studies suggest that priming with an HIV-vaccinia recombinant followed by boosting with subunit envelope proteins offers the most promising strategy to date for a safe and immunogenic vaccine in humans. This study will further examine the combination vaccine approach and define an optimal prime-boost strategy.

DETAILED DESCRIPTION:
Previous studies suggest that priming with an HIV-vaccinia recombinant followed by boosting with subunit envelope proteins offers the most promising strategy to date for a safe and immunogenic vaccine in humans. This study will further examine the combination vaccine approach and define an optimal prime-boost strategy.

Healthy volunteers are randomized to one of eight groups. All patients receive initial immunization with HIVAC-1e, followed by two boosts at months 8 and 12 of rgp120/HIV-1SF2 (BIOCINE), rgp120/HIV-1IIIB (Genentech), rgp120/HIV-1MN (Genentech), or gp160 MN (Immuno-AG). Additionally, half of the patients in each subunit vaccine group receive a repriming with HIVAC-1e at month 4. Subjects are followed for 18 months.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative HIV screening by ELISA, Western blot, and p24 antigen (PBMC HIV culture or HIV-specific PCR can be substituted for Western blot and p24 antigen).
* No history of smallpox (vaccinia) vaccination.
* Normal urinalysis.
* Absolute CD4 count = or > 500 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Subjects with the following conditions are excluded:

* Hepatitis B surface antigenemia.
* Medical or psychiatric condition that precludes compliance with the protocol.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency or chronic illness.
* Eczema within the past year.

Prior Medication:

Excluded:

* Prior experimental HIV vaccine.
* Prior smallpox vaccine.
* Immunoglobulin administration within 2 months prior to enrollment.
* Any experimental agent within 2 months prior to enrollment.
* History of use of immunosuppressive medications.

Prior Treatment:

Excluded:

* Blood or blood product transfusion within the past 6 months.

  1. Current high risk for HIV transmission (persons previously at high risk for HIV transmission can be enrolled provided they have a negative HIV screening and no high-risk behavior has been practiced within the last 6 months).
* Household contact with anyone who is pregnant, has eczema, is less than 12 months of age, or has immunodeficiency disease or is using immunosuppressive medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Study Completion 1994-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Univ. of Rochester AVEG, Rochester, New York
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Clements ML, Corey L, Weinhold K, Schwartz D, Siliciano R, Matthews T, Hsieh R, Graham B, Keefer M, Gorse G, Zolla-Pazner S, Mascola J, Duliege A, Excler J, Tartaglia J, Paoletti E, Hu SL. HIV immunity induced by priming with canarypox or vaccinia-gp160 recombinants and boosting with rgp120. Inst of Hum Virol Annu Meet. 1996 Sept 7-13
- [Background] Corey L, McElrath MJ, Weinhold K, Matthews T, Stablein D, Graham B, Keefer M, Schwartz D, Gorse G. Cytotoxic T cell and neutralizing antibody responses to human immunodeficiency virus type 1 envelope with a combination vaccine regimen. AIDS Vaccine Evaluation Group. J Infect Dis. 1998 Feb;177(2):301-9. doi: 10.1086/514202. PMID 9466515